CLINICAL TRIAL: NCT04851353
Title: Breast Milk as Multiple Sensory Interventions On Infants' Pain and Physiological Distress During Neonatal Screening Procedures
Brief Title: Multiple Sensory Interventions On Infants' Pain and Physiological Distress During Neonatal Screening Procedures
Acronym: MSI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Defense Medical Center, Taiwan (Other)
Responsible Party: Principal Investigator, Hsiang-Yun Lan, Assistant professor, National Defense Medical Center, Taiwan
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Supportive Care
Other Study IDs: 1-106-05-136
Record Dates: First submitted 2021-04-12; First posted 2021-04-20 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Infant Behavior; Pain, Acute; Physiological Stress; Breast Milk
MeSH Terms: conditions — Infant Behavior; Acute Pain | interventions — Smell; Taste

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- GT+VC (Active Comparator): Gentle touch +Verbal comfort
  Interventions: Behavioral: GT+VC
- GT+VC+Smell (Experimental): Gentle touch +Verbal comfort+ Smell breast milk
  Interventions: Behavioral: GT+VC; Behavioral: Smell
- GT+VC+Smell+Taste (Experimental): Gentle touch +Verbal comfort+ Smell breast milk+ Taste milk
  Interventions: Behavioral: GT+VC; Behavioral: Smell; Behavioral: Taste

INTERVENTIONS:
Behavioral: GT+VC — Gentle touch and verbal comfort,
Behavioral: Smell — Smell breast milk
  Arms: GT+VC+Smell; GT+VC+Smell+Taste
Behavioral: Taste — Taste breast milk
  Arms: GT+VC+Smell+Taste

SUMMARY:
The study purposes are to compare the effects of different combinations of sensory interventions on newborns' pain responses, physiological distress (heart rate and oxygen saturation), and crying event during heel stick procedures.

DETAILED DESCRIPTION:
Newborns undergo many necessary invasive procedures for routine care, but these treatments may cause stress and pain. The study purposes are to compare the effects of different combinations of sensory interventions on newborns' pain responses, physiological distress (heart rate and oxygen saturation), and crying event during heel stick procedures. This study was a prospective, randomized controlled trial. Infants were recruited by convenience sampling in a baby room of a medical center in northern Taiwan from September in 2017 to September in 2018. Newborns who met the criteria were recruited by blocked random to three treatment groups: (1)Gentle touch + Verbal comfort, (2) Smell + gentle touch + Verbal comfort, (3) Smell + Taste + Touch + Verbal comfort. Pain response was measured by the Neonatal Infant Pain Scale (NIPS). The physical distress events were measured by the abnormal heart rate and oxygen saturation event, and crying event. All data were collected 5 minutes before heel-stick (baseline), during heel-stick and in recovery status.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age > 36 weeks, birth weight > 2200 g, and at least one parent agreed to participate.

Exclusion Criteria:

* had congenital anomalies and neurologic impairment

Ages: 2 Days to 1 Week | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 250 (Actual)
Dates: Start 2017-09-26 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-09-25 (Actual)

PRIMARY OUTCOMES:
Infants' pain reponse | Six months
  Neonatal Infant Pain Scale

SECONDARY OUTCOMES:
The distress events of physiological parameters | Six months
  Heart rate, oxygen saturation, and crying event

CONTACTS AND LOCATIONS:
Locations (1):
- National defense medical center, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No